CLINICAL TRIAL: NCT03226288
Title: Integrated 3D Surface Scanning System Combined With Soft Tissue and Skeleton Information: Customized Shoe-padding Orthotics for Plantar Fasciitis
Brief Title: Customized Shoe-padding Orthotics for Plantar Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 201704063RIND
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Plantar Fasciitis of Both Feet
Keywords: Plantar Fascitis; orthopedic; 3D surface scanning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While human body receives large external force or motions, minor injuries to the soft tissues will be produced and will lead to acute or chronic inflammation reactions. Plantar fasciitis is the most common foot diseases in normal population. Plantar fascia is a tight band-like soft tissue that crosses between the bony surfaces of the bottom of the foot with thick ligament-like structure substantially. Various reasons will induce the happening of plantar fasciitis including native bone structure, aging, athletic motions and injuries. Indeed, diagnosis of chronic heel pain remains challenging due to the complex structures of the foot. Therefore, it is widely accepted that diagnostic imaging such as ultrasound and computed tomography offer important orthopedic information for clinical assessments of soft tissues and bone. Even though there is no single treatment shows the highest level of evidence for plantar fasciitis, wearing of insoles or orthotics are highly suggested for clinical therapy. Common custom-made insoles are manufactured with polymeric materials based on standing foot-pressure distribution. However, this method strongly depends on experience of doctors or physical therapists and usually time-consuming. In addition, modern medical researches tend to combine the information of both soft (pressure distribution) and hard (orthopedic) tissues for designing of orthotics and other medical assistive devices because of the complicity of the limb motion and structures. Therefore, investigators aim at developing integrated 3D system that provides a 3D limb data model with high-resolution appearance scanning and orthopedic information for designing of medical assistant devices. This model composes of 3D surface scanning, 3D bony structure scanning, and soft tissues characteristic mechanical properties. By developing this system, the 3D model is also highly applicable to the other parts of human assistant devices. It will bring the enormous impact to the associated medical field and create excellent economic value.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old
* Plantar fasciitis patients recommended to use shoe-padding orthotics for treatment

Exclusion Criteria:

* Plantar fasciitis caused by specific reasons, eg. trauma, bone spur, Acute Bursitis.
* Not Taiwanese

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental group: Plantar fasciitis patients recommended to use shoe-padding orthotics for treatment
  Control group: Normal Adults (or without foot disease)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Design customized shoe-padding orthotics for plantar fasciitis | 3 months
  Combine the information of soft (pressure distribution) , hard (orthopedic) tissues and bone (CT) for designing of orthotics

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hao Mike Chang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH East Campus, Research building, Room 946, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided